CLINICAL TRIAL: NCT03113461
Title: Changing the Trajectory of Mild Cognitive Impairment With CPAP Treatment of Obstructive Sleep Apnea
Brief Title: MCI: CPAP Treatment of OSA (Memories2)
Acronym: MCI:OSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PD10057866; R01AG054435 (NIH)
Record Dates: First submitted 2017-04-09; First posted 2017-04-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Mild Cognitive Impairment; Sleep Apnea, Obstructive
Keywords: cognitive impairment; sleep apnea; positive airway pressure therapy
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: CPAP intervention
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- CPAP adherent (Experimental): Study participants in this arm are using the CPAP intervention consistently
  Interventions: Device: CPAP
- CPAP non-adherent (Active Comparator): Study participants in this arm are not using the CPAP intervention consistently
  Interventions: Device: CPAP
- No OSA (No Intervention): Study participants who do not have OSA

INTERVENTIONS:
Device: CPAP — non-invasive positive airway pressure applied using an oronasal mask
  Other Names: continuous positive airway pressure therapy
  Arms: CPAP adherent; CPAP non-adherent

SUMMARY:
The purpose of this project is to determine whether obstructive sleep apnea (OSA) treatment with positive airway pressure therapy (CPAP) can delay the progression of cognitive impairment in patients with amnestic Mild Cognitive Impairment (MCI) as measured by cognitive testing, and brain magnetic resonance imaging (MRI) scans. Study participants will be assessed at baseline, six-month (cognitive tests only) and one-year follow-up.

DETAILED DESCRIPTION:
A growing number of research studies suggest that obstructive sleep apnea (OSA), characterized by episodic nocturnal collapse of the upper airway and reduction/cessation of breathing leading to significant nocturnal hypoxia, is associated with an increased risk of cognitive impairment. OSA is effectively treated with continuous positive airway pressure (CPAP), a pressurized nasal/face mask worn during sleep, but health care providers do not often prescribe it for Mild Cognitive Impairment (MCI) because there are no large, prospective research studies in this population confirming efficacy.

This multi-site study will have a sample size of n=460 divided into three groups followed for one year: 1) a CPAP adherent group (approximately n=200); 2) two control groups consisting of 2a) a CPAP non-adherent control group (approximately n=160) and 2b) a no apnea control group (n=100). This will allow us to confirm whether CPAP treatment, controlling for risk factors such as neuroimaging findings and OSA severity at baseline, predicts the primary outcome of cognitive function at 1-year follow-up. Study participants will also undergo an Amyloid PET scan, use wearable activity monitors and functional/structural MRI brain scans.

This research study will thus examine the one year effects of CPAP on cognitive function and elucidate physiological mechanisms for cognitive decline in aMCI and OSA.

ELIGIBILITY:
Inclusion Criteria:

1. age 55-85 years;
2. moderate to severe OSA as defined by an AHI ≥ 15 events/hr, or no apnea defined by an AHI<5 events/hr using American Academy of Sleep Medicine (AASM) diagnostic methodology as determined on a diagnostic polysomnography;
3. Scoring education adjusted scores 28-35 (inclusive) on optional Telephone Interview for Cognitive Status Modified (pre-screen);
4. Scoring 0-0.5 on the Clinical Dementia Rating Scale (CDR);
5. Scoring 23-30 on the Mini Mental State Examination (MMSE) (exceptions may be made for participants with <8 years of education as determined by the clinical research team);
6. Memory impairment approximately 1.0-1.5 standard deviations below normal (adjusted for age and education) determined by scores on the Logical Memory II a test from the Wechsler memory scale;
7. permitted medications (antidepressants, etc.) stable for at least 4 weeks (12 weeks for cholinesterase inhibitors/memantine) as per ADNI3 criteria;
8. Non-depressed: Scoring < 6 on the Geriatric Depression Scale;
9. study partner, defined as an informant/caregiver who will be able to answer questions about the study participant, and meets one of the following criteria: (a) lives with the participant; (b) spends at least 3 times per week in-person contact with the participant; (c) spends at least 3 times per week in phone contact with the participant; or (d) spends at least 10 hours per week in any combination of phone or in person contact;
10. adequate visual and auditory acuity to allow testing;
11. Post-menopause or surgically sterile;
12. testability - willing and able to complete baseline, 6-month, and 1-year outcome measures, and willing to send in the CPAP Smartcard for adherence;
13. completed at least 6 grades of education; and
14. fluent in English or Spanish.

Exclusion Criteria:

1. any significant neurologic disease other than aMCI, such as Parkinson's Disease, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, multiple sclerosis, head trauma followed by permanent neurologic deficits or known congenital brain structure abnormalities; within the past 6 months brain tumor, or seizure disorder, or subdural hematoma, or post-stroke (based on Modified Hachinski Ischemic Score);
2. Optional: MRI exclusions - presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body; however, the participant has the option of participating in the study without having an MRI;
3. psychiatric disorders, including uncontrolled major depression, newly diagnosed or exacerbation in past 6 months of bipolar disorder as described in the DSM-IV, psychotic features, agitation or behavioral problems within the past 6 months that could lead to difficulty complying with the protocol, or history of schizophrenia (DSM-IV criteria);
4. history of alcohol abuse or dependence within the past 6 months (DSM-IV criteria);
5. any current significant systemic illness or unstable medical condition that could lead to difficulty in complying with the protocol (such as unstable cardiovascular disease); current use of supplemental oxygen or hypoxemia indicated by documented daytime oxyhemoglobin saturation <90% on room air, uncontrolled thyroid disease (to be included must be on stable dose of thyroid medication for >6 months), uncontrolled cirrhosis, cancer diagnosis within the past 6 months (exceptions may be made at the PI's discretion depending on cancer severity and the treatment required), clinically significant laboratory abnormalities such as reported untreated folate, B12, or TSH disease, or resident of a skilled nursing facility;
6. participation in clinical studies involving neuropsychological measures being conducted more than twice a year;
7. received and was adherent to CPAP or bi-level pressure for OSA within the past 6 months;

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Digit Symbol-Coding test | one-year follow-up
  incorporates both elements of memory and processing speed and correlates with executive functioning

SECONDARY OUTCOMES:
Clinical Dementia Rating Scale | one-year follow-up
  Assessment of global cognition

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka Gooneratne, MD, MSc, Principal Investigator — Associate Professor; Kathy Richards, PhD, Principal Investigator — Professor; David Wolk, MD, Principal Investigator — Associate Professor
Locations (4):
- United States (4):
  - Washington University in St. Louis, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Pending